CLINICAL TRIAL: NCT03965923
Title: Phase 3b, Randomized, Open Label Safety Trial of Dapivirine Vaginal Ring and Oral TRUVADA® Use in Pregnancy
Brief Title: Randomized, Open Label Safety Trial of Dapivirine Vaginal Ring and Oral TRUVADA® Use in Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: MTN-042; 38544 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Dapivirine; Contraceptive Devices, Female; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Cohort 1 Mothers: Dapivirine (DPV) Vaginal Ring (VR) (Experimental): Participants in Cohort 1 (36 0/7 weeks - 37 6/7 weeks) will use one DPV VR continuously for approximately one month, replacing the DPV VR each month. Participants will use the DPV VR until their pregnancy outcome but no later than 41 6/7 weeks of gestation.
  Interventions: Drug: Dapivirine (DPV) Vaginal Ring (VR)
- Cohort 1 Mothers: Truvada Tablet (Experimental): Participants in Cohort 1 (36 0/7 weeks - 37 6/7 weeks) will take one Truvada oral tablet daily. Participants will take Truvada until their pregnancy outcome but no later than 41 6/7 weeks of gestation.
  Interventions: Drug: Truvada Tablet
- Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) (Experimental): Participants in Cohort 2 (30 0/7 weeks - 35 6/7 weeks) will use one DPV VR continuously for approximately one month, replacing the DPV VR each month. Participants will use the DPV VR until their pregnancy outcome but no later than 41 6/7 weeks of gestation.
  Interventions: Drug: Dapivirine (DPV) Vaginal Ring (VR)
- Cohort 2 Mothers: Truvada Tablet (Experimental): Participants in Cohort 2 (30 0/7 weeks - 35 6/7 weeks) will take one Truvada oral tablet daily. Participants will take Truvada until their pregnancy outcome but no later than 41 6/7 weeks of gestation.
  Interventions: Drug: Truvada Tablet
- Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR) (Experimental): Participants in Cohort 3 (12 0/7 weeks - 29 6/7 weeks) will use one DPV VR continuously for approximately one month, replacing the DPV VR each month. Participants will use the DPV VR until their pregnancy outcome but no later than 41 6/7 weeks of gestation.
  Interventions: Drug: Dapivirine (DPV) Vaginal Ring (VR)
- Cohort 3 Mothers: Truvada Tablet (Experimental): Participants in Cohort 3 (12 0/7 weeks - 29 6/7 weeks) will take one Truvada oral tablet daily. Participants will take Truvada until their pregnancy outcome but no later than 41 6/7 weeks of gestation.
  Interventions: Drug: Truvada Tablet
- Cohort 1 Infants: Dapivirine (DPV) Vaginal Ring (VR) (Experimental): Infants born to maternal participants in the Cohort 1 (36 0/7 weeks - 37 6/7 weeks) DPV VR arm.
  Interventions: Drug: Dapivirine (DPV) Vaginal Ring (VR)
- Cohort 1 Infants: Truvada Tablet (Experimental): Infants born to maternal participants in the Cohort 1 (36 0/7 weeks - 37 6/7 weeks) Truvada oral tablet daily arm.
  Interventions: Drug: Truvada Tablet
- Cohort 2 Infants: Dapivirine (DPV) Vaginal Ring (VR) (Experimental): Infants born to maternal participants in the Cohort 2 (30 0/7 weeks - 35 6/7 weeks) DPV VR arm.
  Interventions: Drug: Dapivirine (DPV) Vaginal Ring (VR)
- Cohort 2 Infants: Truvada Tablet (Experimental): Infants born to maternal participants in the Cohort 2 (30 0/7 weeks - 35 6/7 weeks) Truvada oral tablet daily arm.
  Interventions: Drug: Truvada Tablet
- Cohort 3 Infants: Dapivirine (DPV) Vaginal Ring (VR) (Experimental): Infants born to maternal participants in the Cohort 3 (12 0/7 weeks - 29 6/7 weeks) DPV VR arm.
  Interventions: Drug: Dapivirine (DPV) Vaginal Ring (VR)
- Cohort 3 Infants: Truvada Tablet (Experimental): Infants born to maternal participants in the Cohort 3 (12 0/7 weeks - 29 6/7 weeks) Truvada oral tablet daily arm.
  Interventions: Drug: Truvada Tablet

INTERVENTIONS:
Drug: Dapivirine (DPV) Vaginal Ring (VR) — Vaginal ring containing 25 mg of DPV
  Arms: Cohort 1 Infants: Dapivirine (DPV) Vaginal Ring (VR); Cohort 1 Mothers: Dapivirine (DPV) Vaginal Ring (VR); Cohort 2 Infants: Dapivirine (DPV) Vaginal Ring (VR); Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR); Cohort 3 Infants: Dapivirine (DPV) Vaginal Ring (VR); Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR)
Drug: Truvada Tablet — Tablet taken orally
  Other Names: Emtricitabine/Tenofovir Disoproxil Fumarate; FTC/TDF
  Arms: Cohort 1 Infants: Truvada Tablet; Cohort 1 Mothers: Truvada Tablet; Cohort 2 Infants: Truvada Tablet; Cohort 2 Mothers: Truvada Tablet; Cohort 3 Infants: Truvada Tablet; Cohort 3 Mothers: Truvada Tablet

SUMMARY:
The purpose of this study is to evaluate the maternal and infant safety of the dapivirine (DPV) vaginal ring (VR) and daily oral Truvada in HIV-uninfected pregnant women and their infants.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the maternal and infant safety of the dapivirine (DPV) vaginal ring (VR) and daily oral Truvada in HIV-uninfected pregnant women and their infants.

Participants will be assigned to one of three cohorts based on gestational age:

* Cohort 1: 36 0/7 weeks - 37 6/7 weeks
* Cohort 2: 30 0/7 weeks - 35 6/7 weeks
* Cohort 3: 12 0/7 weeks - 29 6/7 weeks

Within each cohort, participants will be randomized to receive either DPV VR or oral Truvada. Participants randomized to the DPV VR will use the VR continuously for approximately one month, replacing the VR each month. Participants taking the Truvada tablet will take one tablet orally per day. Participants will use their assigned study product until their pregnancy outcome, but no later than 41 6/7 weeks of gestation.

Participants will attend several study visits throughout the study and study staff will also contact participants by phone at different timepoints throughout the study.

The total duration of study participation will vary depending on gestational age at time of enrollment and length of pregnancy prior to pregnancy outcome and will range from approximately 12 weeks or less for Cohort 1 to approximately 36 weeks or less for Cohort 3. Infants born to study participants will be followed for approximately 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 40 years (inclusive) at Enrollment, verified per site standard operating procedures (SOPs).
* At Enrollment, evidence of a viable, intrauterine, singleton pregnancy with sonographic confirmation, including for gestational age assessment.

  * Note: If adequate (per judgment of Investigator of Record [IoR]/designee) sonographic results are not available from medical records at Screening, an ultrasound must be performed and results be available for review at Enrollment for all Cohorts. The ultrasound should be performed no later than the 36th week of gestation for Cohort 1 or the 28th week of gestation for Cohort 2.
* At Enrollment, pregnancy within gestational age limits of the currently enrolling cohort (per the study protocol).
* HIV-uninfected based on testing performed at Screening and Enrollment (per protocol algorithm in the study protocol).
* At Screening and Enrollment, intending to continue her pregnancy until delivery.
* At Screening and Enrollment, intending to deliver at a health center or hospital where adequate records may be obtained, as defined in site SOPs.

  * Note: Plans to deliver at a health center or hospital where adequate records may be obtained is inclusionary due to logistical challenges related to collection of vaginal rings (VRs), specimens and delivery outcome data outside of those settings.
* At Screening and Enrollment, willing to be randomized at time of enrollment to either of the two study arms, and to continue study product use until delivery.
* Able and willing to comply with all study requirements and complete all study procedures.
* Able and willing to provide the following:

  * Informed consent for her and her infant to be screened for and to enroll in MTN-042, as defined in site SOPs.
  * Adequate locator information, as defined in site SOPs.
  * Adequate documentation of registration for antenatal care, as defined in site SOPs.
  * Permission to contact participant's antenatal and postpartum care provider(s) and to obtain copies of antenatal and postpartum care records.
* At Screening and Enrollment, agrees not to participate in other research studies involving drugs, medical devices, vaginal products, or vaccines for the duration of study participation, unless approved by the Protocol Safety Review Team (PSRT).

Exclusion Criteria:

* Per participant report at Screening and/or Enrollment, intends to do any of the following during the study participation period:

  * Use oral pre-exposure prophylaxis (PrEP) outside the context of study participation.
  * Relocate away from the study site.
  * Travel away from the study site for a time period that would interfere with study participation.
* At Screening or Enrollment, has a positive HIV test.
* At Screening or Enrollment, diagnosed with urinary tract infection (UTI), cervicitis, sexually transmitted infection (STI) or reproductive tract infection (RTI) requiring treatment per World Health Organization (WHO) guidelines.

  * Note: Detection of bacterial vaginosis (BV) or candida in the absence of symptoms is not exclusionary. Otherwise eligible participants diagnosed during screening with a UTI, cervicitis, or STI/RTI requiring treatment per WHO guidelines are offered treatment consistent with WHO recommendations. If treatment is completed and symptoms have resolved within 35 days of obtaining informed consent for screening, the participant may be enrolled.
* At Enrollment, has a clinically apparent Grade 2 or higher pelvic exam finding.*

  * Note: Cervical friability bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the Investigator of Record (IoR)/designee is considered expected bleeding and is not exclusionary.
* Participant report, clinical evidence and/or antenatal/medical care record of any of the following:

  * Currently breastfeeding at Enrollment.
  * Known adverse reaction to any of the study products (ever).
  * Known adverse reaction to latex and polyurethane (ever).
  * Symptoms suggestive of acute HIV infection at Screening or Enrollment.
  * Non-therapeutic injection drug use in the 12 months prior to Enrollment.
  * Use of HIV post-exposure prophylaxis (PEP) and/or PrEP during the current pregnancy.
  * Participation in any other research study involving drugs, medical devices, vaginal products, or vaccines during the current pregnancy.
  * At Screening or Enrollment, known to have any of the following during the current pregnancy:

    * Multiple gestation
    * Placenta previa
    * Cervical cerclage
    * Abnormal fetal anatomy (in the opinion of the IoR or designee)
    * Intrauterine growth restriction
    * Pre-existing or gestational diabetes
    * Hypertensive disorder of pregnancy
    * Severe malaria
    * Treatment for preterm labor
    * Abnormal quantity of amniotic fluid (oligohydramnios or polyhydramnios)
  * At Screening, known to have had any of the following in a previous pregnancy:

    * Intrauterine growth restriction
    * Gestational diabetes
    * Hypertensive disorder of pregnancy
    * Intrauterine fetal demise (estimated gestational age greater than or equal to 20 weeks)
    * Delivery prior to 37 0/7 weeks
  * At Enrollment, as determined by the IoR/designee, has any significant obstetrical complication (e.g., premature rupture of membranes, any abnormal placentation) or uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease that would make study participation unsafe.
* At Screening, has any of the following laboratory abnormalities:

  * Positive for hepatitis B surface antigen (HBsAg).
  * Aspartate aminotransferase (AST) or alanine transaminase (ALT) greater than or equal to Grade 1.**
  * Hemoglobin greater than or equal to Grade 2.**
  * Platelet count greater than or equal to Grade 1.**
  * Creatinine greater than or equal to Grade 1.**
  * Estimated creatinine clearance greater than or equal to Grade 2 (Cockcroft Gault formula).**
  * Glycosuria greater than or equal to Grade 2.**
  * Proteinuria greater than or equal to Grade 2.**
  * Note: Otherwise eligible participants with an exclusionary test (other than HBsAg) may be re-tested during the screening process; re-testing procedure details can be found in the MTN-042 Study Specific Procedures (SSP) Manual. If improvement to a non-exclusionary grade or resolution is documented within 35 days of providing informed consent for screening, the participant may be enrolled.
* Has any condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
* *Female Genital Grading Table for Use in Microbicide Studies Addendum 1 (Dated November 2007) to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017.
* **DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1, July 2017.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1104 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bunge, MD, MPH, Study Chair — University of Pittsburgh; Felix Mhlanga, MBChB, MMed, Study Chair — Zengeza Clinical Research Site; Lee Fairlie, Study Chair — Wits RHI Shandukani Research Centre
Locations (4):
- Blantyre CRS (Johns Hopkins Research Project/College of Medicine), Blantyre, Malawi
- Wits RHI Shandukani Research Centre CRS, Johannesburg, Gauteng, South Africa
- MU-JHU Research Collaboration (MUJHU CARE LTD) CRS, Kampala, Uganda
- Zengeza CRS, Chitungwiza, Mashonaland East Province, Zimbabwe

REFERENCES:
- [Derived] Fairlie L, Szydlo DW, Mayo A, Bunge K, Mhlanga F, Piper J, Dadabhai S, Gatsi VM, Horne E, Ssemambo PK, Mandiwa V, Mgodi NM, Owor M, Anderson PL, Marzinke MA, Nakabiito C, Scheckter R, Chappell C, Hillier SL; MTN-042 study team. Safety outcomes among infants whose mothers used the dapivirine vaginal ring or oral PrEP during pregnancy (MTN-042/DELIVER): a randomised phase 3b study. Lancet HIV. 2025 Nov;12(11):e763-e773. doi: 10.1016/S2352-3018(25)00261-9. PMID 41173578
- [Derived] Nansimbe J, Mirembe BG, Ssemambo PK, Ssekasi AM, Byogero R, Nalwoga J, Nakabiito C. Exploring pregnant women's experiences with dapivirine vaginal ring insertion during the MTN-042/DELIVER study in Uganda: a description of secondary data. Ther Adv Infect Dis. 2025 Apr 11;12:20499361251332750. doi: 10.1177/20499361251332750. eCollection 2025 Jan-Dec. PMID 40292084

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 1 Mothers: Truvada Tablet | Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Mothers: Truvada Tablet | Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Mothers: Truvada Tablet | Cohort 1 Infants: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 1 Infants: Truvada Tablet | Cohort 2 Infants: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Infants: Truvada Tablet | Cohort 3 Infants: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Infants: Truvada Tablet
Started | 101 | 49 | 106 | 51 | 202 | 49 | 99 | 48 | 103 | 51 | 197 | 48
Completed | 98 | 46 | 102 | 49 | 198 | 48 | 93 | 43 | 95 | 49 | 189 | 48
Not Completed | 3 | 3 | 4 | 2 | 4 | 1 | 6 | 5 | 8 | 2 | 8 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 3 | 1 | 2 | 0 | 4 | 3 | 4 | 0 | 2 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1 | 0 | 2 | 1 | 2 | 1 | 0 | 2 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 4 | 0
Not completed — Other reason | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 1 Mothers: Truvada Tablet | Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Mothers: Truvada Tablet | Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Mothers: Truvada Tablet | Cohort 1 Infants: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 1 Infants: Truvada Tablet | Cohort 2 Infants: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Infants: Truvada Tablet | Cohort 3 Infants: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Infants: Truvada Tablet | Total
Number analyzed (Participants) | 101 | 49 | 106 | 51 | 202 | 49 | 99 | 48 | 103 | 51 | 197 | 48 | 1104
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Infants were enrolled on their date of birth, so their age in years at enrollment was 0 years by definition and is omitted. Their gestational age at birth is reported as a separate baseline measure.
  years
    number analyzed (Participants) | 101 | 49 | 106 | 51 | 202 | 49 | 0 | 0 | 0 | 0 | 0 | 0 | 558
    (all) | 25.4 (5.4) | 25.1 (5.4) | 26.2 (5.5) | 26.7 (6.2) | 25.7 (5.4) | 24.0 (5.1) |  |  |  |  |  |  | 25.6 (5.5)
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Infant gestational age at birth Population: Infants were enrolled on their date of birth, so their age at enrollment was 0 years by definition. In place of age at enrollment, gestational age at birth is reported. This measure is only collected for infants.
  weeks
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 99 | 48 | 103 | 51 | 197 | 48 | 546
    (all) |  |  |  |  |  |  | 40.1 (1.6) | 39.6 (1.6) | 39.6 (1.8) | 39.4 (1.7) | 39.8 (1.6) | 39.4 (1.5) | 39.7 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The infant analysis population is enrolled infants whose sex at birth was available.
  Participants
    number analyzed (Participants) | 101 | 49 | 106 | 51 | 202 | 49 | 99 | 48 | 103 | 50 | 197 | 48 | 1103
    Female | 101 | 49 | 106 | 51 | 202 | 49 | 48 | 24 | 62 | 24 | 104 | 25 | 845
    Male | 0 | 0 | 0 | 0 | 0 | 0 | 51 | 24 | 41 | 26 | 93 | 23 | 258
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 101 | 49 | 106 | 51 | 202 | 49 | 99 | 48 | 103 | 51 | 197 | 48 | 1104
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Malawi | 18 | 9 | 26 | 14 | 53 | 13 | 18 | 9 | 26 | 13 | 53 | 13 | 265
  South Africa | 28 | 14 | 20 | 8 | 35 | 9 | 26 | 14 | 18 | 8 | 32 | 8 | 220
  Uganda | 30 | 14 | 28 | 14 | 55 | 13 | 30 | 14 | 27 | 15 | 54 | 13 | 307
  Zimbabwe | 25 | 12 | 32 | 15 | 59 | 14 | 25 | 11 | 32 | 15 | 58 | 14 | 312

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Composite Safety Endpoint Adverse Event (AE)
Description: All AEs were reported as per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events. Composite safety endpoint AEs were AEs that were either categorized as serious adverse events (SAEs) or were Grade 3 or higher.
  This measure is the number of participants with at least one composite AE.
Time Frame: Measured through participant's last study visit. For mothers, this occurred at approximately Week 12 to 36, depending on participant's cohort, and for infants at approximately Week 52.
Population: All mothers who were randomized and enrolled are included. All enrolled infants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 1 Mothers: Truvada Tablet | Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Mothers: Truvada Tablet | Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Mothers: Truvada Tablet | Cohort 1 Infants: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 1 Infants: Truvada Tablet | Cohort 2 Infants: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Infants: Truvada Tablet | Cohort 3 Infants: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Infants: Truvada Tablet
Number analyzed (Participants) | 101 | 49 | 106 | 51 | 202 | 49 | 99 | 48 | 103 | 51 | 197 | 48
Participants | 2 | 6 | 16 | 5 | 24 | 4 | 23 | 15 | 30 | 10 | 48 | 6

2. Primary Outcome: Pregnancy Outcomes
Description: Frequency of different types of pregnancy outcomes among mothers.
Time Frame: Measured through participant's last study visit, at approximately Week 12 to 36, depending on participant's cohort
Population: The analysis population is all randomized and enrolled participants with an obtainable pregnancy outcome. The number of units analyzed is the number of pregnancy outcomes, due to the potential for participants to have non-singleton pregnancies.
Measure: Count of Units; unit: Obtainable pregnancy outcomes
Units Other Than Participants: Obtainable pregnancy outcomes
Arm/Group | Cohort 1 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 1 Mothers: Truvada Tablet | Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Mothers: Truvada Tablet | Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Mothers: Truvada Tablet
Number analyzed (Participants) | 99 | 49 | 104 | 50 | 199 | 48
Number analyzed (Obtainable pregnancy outcomes) | 99 | 49 | 104 | 51 | 199 | 48
Obtainable pregnancy outcomes
  Full term live birth (>= 37 0/7 weeks) | 98 | 45 | 97 | 46 | 188 | 45
  Premature live birth (<37 0/7 weeks) | 1 | 3 | 6 | 5 | 8 | 3
  Stillbirth/intrauterine fetal demise (>= 20 0/7 weeks) | 0 | 1 | 1 | 0 | 2 | 0
  Spontaneous abortion (<20 0/7 weeks) | 0 | 0 | 0 | 0 | 1 | 0

3. Secondary Outcome: Pregnancy Complications: Frequency of Pregnancy Complications
Description: Frequency of different types of pregnancy complications among mothers.
  The categories of pregnancy complications were pre-defined on the case report form, and after the completion of Cohort 1 follow-up there were some changes made to the pregnancy complication categories. In Cohort 1 the category "peripartum hemorrhage" was collected, but in Cohort 2 and 3 this category was removed from the list of pre-defined complications. Two other categories, "antepartum hemorrhage" and "intrapartum hemorrhage", were added to the list for Cohort 2 and Cohort 3. As a result, participants in Cohort 1 were not evaluated for antepartum or intrapartum hemorrhage, while participants in Cohorts 2 and 3 were not evaluated for peripartum hemorrhage. All other complications were collected for all three cohorts, and participants in all three cohorts were evaluated for each complication.
Time Frame: Measured through participant's last study visit, at approximately Week 12 to 36, depending on participant's cohort
Population: as for outcome 2
Measure: Count of Units; unit: Obtainable pregnancy outcomes
Units Other Than Participants: Obtainable pregnancy outcomes
Arm/Group | Cohort 1 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 1 Mothers: Truvada Tablet | Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Mothers: Truvada Tablet | Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Mothers: Truvada Tablet
Number analyzed (Participants) | 99 | 49 | 104 | 50 | 199 | 48
Number analyzed (Obtainable pregnancy outcomes) | 99 | 49 | 104 | 51 | 199 | 48
Obtainable pregnancy outcomes
  Hypertensive disorders of pregnancy: Yes | 3 | 4 | 9 | 7 | 20 | 7
  Hypertensive disorders of pregnancy: No | 96 | 45 | 95 | 44 | 179 | 41
  Chronic hypertensive disorder: Yes | 0 | 0 | 0 | 0 | 1 | 0
  Chronic hypertensive disorder: No | 99 | 49 | 104 | 51 | 198 | 48
  Gestational hypertensive disorder: Yes | 3 | 2 | 5 | 7 | 16 | 6
  Gestational hypertensive disorder: No | 96 | 47 | 99 | 44 | 183 | 42
  Pre-eclampsia without severe features: Yes | 0 | 1 | 1 | 0 | 3 | 0
  Pre-eclampsia without severe features: No | 99 | 48 | 103 | 51 | 196 | 48
  Pre-eclampsia with severe features: Yes | 0 | 1 | 2 | 0 | 1 | 1
  Pre-eclampsia with severe features: No | 99 | 48 | 102 | 51 | 198 | 47
  Eclampsia: Yes | 0 | 0 | 0 | 0 | 0 | 0
  Eclampsia: No | 99 | 49 | 104 | 51 | 199 | 48
  Unspecified hypertensive disorder: Yes | 0 | 0 | 1 | 0 | 0 | 0
  Unspecified hypertensive disorder: No | 99 | 49 | 103 | 51 | 199 | 48
  Chorioamnionitis: Yes | 0 | 0 | 1 | 0 | 0 | 0
  Chorioamnionitis: No | 99 | 49 | 103 | 51 | 199 | 48
  Puerperal sepsis: Yes | 0 | 0 | 0 | 2 | 0 | 0
  Puerperal sepsis: No | 99 | 49 | 104 | 49 | 199 | 48
  Endometritis: Yes | 0 | 0 | 0 | 1 | 0 | 0
  Endometritis: No | 99 | 49 | 104 | 50 | 199 | 48
  Peripartum hemorrhage: number analyzed (Participants) | 99 | 49 | 0 | 0 | 0 | 0
  Peripartum hemorrhage: number analyzed (Obtainable pregnancy outcomes) | 99 | 49 | 0 | 0 | 0 | 0
  Peripartum hemorrhage: Yes | 2 | 1 | 0 | 0 | 0 | 0
  Peripartum hemorrhage: No | 97 | 48 | 0 | 0 | 0 | 0
  Antepartum hemorrhage: number analyzed (Participants) | 0 | 0 | 104 | 50 | 199 | 48
  Antepartum hemorrhage: number analyzed (Obtainable pregnancy outcomes) | 0 | 0 | 104 | 51 | 199 | 48
  Antepartum hemorrhage: Yes | 0 | 0 | 2 | 1 | 2 | 0
  Antepartum hemorrhage: No | 0 | 0 | 102 | 50 | 197 | 48
  Intrapartum hemorrhage: number analyzed (Participants) | 0 | 0 | 104 | 50 | 199 | 48
  Intrapartum hemorrhage: number analyzed (Obtainable pregnancy outcomes) | 0 | 0 | 104 | 51 | 199 | 48
  Intrapartum hemorrhage: Yes | 0 | 0 | 0 | 1 | 3 | 0
  Intrapartum hemorrhage: No | 0 | 0 | 104 | 50 | 196 | 48
  Postpartum hemorrhage: Yes | 2 | 1 | 2 | 0 | 4 | 0
  Postpartum hemorrhage: No | 97 | 48 | 102 | 51 | 195 | 48
  Preterm premature rupture of membranes (PPROM): Yes | 0 | 0 | 1 | 0 | 3 | 0
  Preterm premature rupture of membranes (PPROM): No | 99 | 49 | 103 | 51 | 196 | 48
  Fever of unclear etiology: Yes | 0 | 0 | 0 | 0 | 0 | 0
  Fever of unclear etiology: No | 99 | 49 | 104 | 51 | 199 | 48
  Other complication: Yes | 1 | 1 | 4 | 0 | 2 | 1
  Other complication: No | 98 | 48 | 100 | 51 | 197 | 47

4. Secondary Outcome: Infant Drug Levels: Number of Infants With Detectable Infant Blood Tenofovir Diphosphate (TFV-DP)
Description: Infant blood TFV-DP was measured at infants' post pregnancy outcome (PPO) visit (up to 14 days after pregnancy outcome). The outcome is defined as having detectable drug level, with detectable drug levels defined as a TFV-DP concentration above the lower limit of quantification (LLOQ) for the assay.
Time Frame: Measured at the 2-week post pregnancy outcome (PPO) visit
Population: Enrolled infants with an analyzable sample collected at the PPO visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Infants: Truvada Tablet | Cohort 2 Infants: Truvada Tablet | Cohort 3 Infants: Truvada Tablet
Number analyzed (Participants) | 44 | 50 | 43
Participants | 30 | 35 | 30

5. Secondary Outcome: Infant Drug Levels: Number of Infants With Detectable Blood Emtricitabine Triphosphate (FTC-TP)
Description: Infant blood FTC-TP was measured at infants' PPO visit. The outcome is defined as having detectable drug level, with detectable drug levels defined as a FTC-TP concentration above the lower limit of quantification (LLOQ) for the assay.
Time Frame: measured at the 2-week post pregnancy outcome (PPO) visit
Population: Enrolled infants with an analyzable sample collected at the PPO visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Infants: Truvada Tablet | Cohort 2 Infants: Truvada Tablet | Cohort 3 Infants: Truvada Tablet
Number analyzed (Participants) | 44 | 50 | 43
Participants | 7 | 6 | 1

6. Secondary Outcome: Infant Drug Levels: Number of Infants With Detectable Plasma DPV
Description: Infant plasma DPV concentration was measured at infants' post pregnancy outcome (PPO) visit (up to 14 days after pregnancy outcome). The outcome is defined as having detectable drug level, with detectable drug levels defined as a DPV concentration above the lower limit of quantification (LLOQ) for the assay.
Time Frame: measured at the 2-week post pregnancy outcome (PPO) visit
Population: Enrolled infants with an analyzable sample collected at the PPO visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Infants: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Infants: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Infants: Dapivirine (DPV) Vaginal Ring (VR)
Number analyzed (Participants) | 94 | 97 | 182
Participants | 22 | 31 | 30

7. Secondary Outcome: Adherence: Maternal Blood TFV-DP Concentrations
Description: Maternal blood TFV-DP was collected at the 2-week, bi-weekly (starting at 4-weeks), and PPO visits for participants randomized to receive Truvada Tablet. In Cohort 1 this was done for a randomly selected subset of those participants. Participants are categorized as ever being exposed if they had at least one measure that was >= 200 fmol/punch (if the sample was collected more than 6 weeks after randomization) or >= 150 fmol/punch (if the sample was collected within 6 weeks of randomization). They are categorized as never being exposed if they had at least one analyzable sample and none met the criteria.
Time Frame: Measured through participant's 2-week PPO visit, at approximately Week 8-32, depending on participant's cohort
Population: Participants enrolled and randomized to the Truvada Tablet arm who had at least one analyzable blood TFV-DP sample collected during study follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Mothers: Truvada Tablet | Cohort 2 Mothers: Truvada Tablet | Cohort 3 Mothers: Truvada Tablet
Number analyzed (Participants) | 15 | 51 | 49
Participants
  Ever exposed | 8 | 37 | 41
  Never exposed | 7 | 14 | 8

8. Secondary Outcome: Adherence: Maternal Blood FTC-TP Concentrations
Description: Maternal blood FTC-TP was collected at the 2-week, bi-weekly (starting at 4-weeks), and PPO visits for participants randomized to receive Truvada Tablet. In Cohort 1 this was done for a randomly selected subset of those participants.
Time Frame: Measured through participant's 2-week PPO visit, at approximately Week 8-32, depending on participant's cohort
Population: Participants enrolled and randomized to the Truvada Tablet arm who had an analyzable blood FTC-TP sample collected during at their PPO visit.
Measure: Mean (Standard Deviation); unit: pmol
Arm/Group | Cohort 1 Mothers: Truvada Tablet | Cohort 2 Mothers: Truvada Tablet | Cohort 3 Mothers: Truvada Tablet
Number analyzed (Participants) | 14 | 47 | 45
pmol | 0.1 (0.2) | 0 (0) | 0 (0)

9. Secondary Outcome: Adherence: Maternal Plasma DPV Concentrations
Description: Maternal plasma DPV was collected at the 2-week, bi-weekly (starting at 4-weeks), and PPO visits for a randomly selected subset of participants (approximately 50%) randomized to receive the VR. Participants are categorized as ever being exposed if they had at least one measure that was greater than the LLOQ (i.e., greater than or equal to 20 pg/mL). They are categorized as never being exposed if they had at least one analyzable sample and none met the criteria.
Time Frame: Measured through participant's 2-week PPO visit, at approximately Week 8-32, depending on participant's cohort
Population: Participants enrolled and randomized to the VR arm who had at least one analyzable plasma DPV sample collected during study follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR)
Number analyzed (Participants) | 48 | 52 | 100
Participants | 43 | 51 | 98

10. Secondary Outcome: Adherence: Frequency of Missing Taking the Pills
Description: Based on participant report, as defined by self-reported missed doses for oral Truvada. This was only reported by participants in Cohorts 2 and 3.
Time Frame: Measured at Week 4 and PPO visits
Population: Participants enrolled and randomized to the Truvada Tablet arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 Mothers: Truvada Tablet | Cohort 3 Mothers: Truvada Tablet
Number analyzed (Participants) | 51 | 49
Participants
  Week 4 Visit: Never | 36 | 35
  Week 4 Visit: Rarely | 8 | 11
  Week 4 Visit: Often | 0 | 0
  Week 4 Visit: Missing | 7 | 3
  PPO Visit: Never | 39 | 35
  PPO Visit: Rarely | 6 | 10
  PPO Visit: Often | 2 | 0
  PPO Visit: Missing | 4 | 4

11. Secondary Outcome: Adherence: Number of Participants With Product Exposure (Measured in Residual Drug Levels in Returned VRs)
Description: Residual drug levels were collected from returned VRs, which were expected to be returned at monthly visits throughout study follow-up. Drug release rate was calculated by subtracting the residual level from the amount of residual drug in the manufacturer lot, divided by the number of days the participant was expected to use that ring, times 28 days. For each individual ring, a ring was considered to show evidence of use if the residual drug level was greater than or equal to 0.9mg/28 days of use.
  Participants are categorized as either ever being exposed or never being exposed to product over the course of study follow-up. They are categorized as ever being exposed to product if they had at least one ring with evidence of use (i.e., greater than or equal to 0.9 mg/28 days of release). They are categorized as never being exposed if they had at least one analyzable returned ring and none of these rings had evidence of use.
Time Frame: Measured through participant's last study visit, at approximately Week 12 to 36, depending on participant's cohort
Population: Participants enrolled and randomized to the VR arm who had at least one analyzable residual drug level collected during study follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR)
Number analyzed (Participants) | 97 | 105 | 199
Participants | 95 | 93 | 193

12. Secondary Outcome: Acceptability: Participant Willingness to Use Study Products During Pregnancy in the Future
Description: Based on participant report of whether they would be willing to use the study product they were randomized to receive when pregnant in the future. Only asked of participants in Cohorts 2 and 3.
Time Frame: Measured at Week 4 and 6-Week PPO/SEV visits.
Population: Participants enrolled and randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Mothers: Truvada Tablet | Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Mothers: Truvada Tablet
Number analyzed (Participants) | 106 | 51 | 199 | 49
Participants
  Week 4 Visit: Yes | 98 | 42 | 193 | 49
  Week 4 Visit: No | 0 | 2 | 3 | 0
  Week 4 Visit: Not sure | 3 | 1 | 2 | 0
  Week 4 Visit: N/A: doesn't plan to have future pregnancies | 2 | 0 | 0 | 0
  Week 4 Visit: Missing | 3 | 6 | 1 | 0
  6-Week PPO Visit/SEV: Yes | 94 | 46 | 190 | 46
  6-Week PPO Visit/SEV: No | 3 | 0 | 2 | 0
  6-Week PPO Visit/SEV: Not sure | 3 | 1 | 1 | 0
  6-Week PPO Visit/SEV: N/A: doesn't plan to have future pregnancies | 1 | 1 | 0 | 0
  6-Week PPO Visit/SEV: Missing | 5 | 3 | 6 | 3

13. Secondary Outcome: Acceptability: Participants Who Find the Study Products to be at Least as Acceptable as Other HIV Prevention Methods
Description: Based on participant report of how much they liked or disliked the study product they were randomized to receive for HIV prevention, and of how much they liked or disliked male condoms for HIV prevention. Only asked of participants in Cohorts 2 and 3.
Time Frame: Measured at Week 4 visits.
Population: Participants enrolled and randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Mothers: Truvada Tablet | Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Mothers: Truvada Tablet
Number analyzed (Participants) | 106 | 51 | 202 | 49
Participants
  How much do you like or dislike male condoms for HIV prevention: Dislike very much | 23 | 5 | 25 | 7
  How much do you like or dislike male condoms for HIV prevention: Dislike | 30 | 19 | 96 | 23
  How much do you like or dislike male condoms for HIV prevention: Neither like nor dislike | 10 | 8 | 25 | 6
  How much do you like or dislike male condoms for HIV prevention: Like | 28 | 12 | 45 | 11
  How much do you like or dislike male condoms for HIV prevention: Like very much | 12 | 1 | 7 | 2
  How much do you like or dislike male condoms for HIV prevention: Missing | 3 | 6 | 4 | 0
  How much do you like or dislike the [pills/ring] for HIV prevention: Dislike very much | 2 | 0 | 3 | 1
  How much do you like or dislike the [pills/ring] for HIV prevention: Dislike | 2 | 0 | 2 | 0
  How much do you like or dislike the [pills/ring] for HIV prevention: Neither like nor dislike | 1 | 4 | 1 | 2
  How much do you like or dislike the [pills/ring] for HIV prevention: Like | 47 | 29 | 122 | 32
  How much do you like or dislike the [pills/ring] for HIV prevention: Like very much | 51 | 12 | 70 | 14
  How much do you like or dislike the [pills/ring] for HIV prevention: Missing | 3 | 6 | 4 | 0

14. Secondary Outcome: Adherence: Frequency of Ring Removal/Expulsion
Description: Based on participant report, as defined by self-reported occurrences of the ring being out of the vagina for more than 12 hours, being out for any time. This was only reported by participants in Cohorts 2 and 3.
Time Frame: Measured at Week 4 visit and Post-Pregnancy Outcome (PPO) (occurring within 2 weeks of pregnancy outcome) visit
Population: Participants enrolled and randomized to the Truvada Tablet arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR)
Number analyzed (Participants) | 106 | 202
Participants
  Ring out for >12 hours in past 4 weeks - Week 4 Visit: Never | 101 | 190
  Ring out for >12 hours in past 4 weeks - Week 4 Visit: Rarely | 1 | 4
  Ring out for >12 hours in past 4 weeks - Week 4 Visit: Often | 0 | 2
  Ring out for >12 hours in past 4 weeks - Week 4 Visit: Missing | 4 | 6
  Ring out for >12 hours in past 4 weeks - PPO Visit: Never | 93 | 145
  Ring out for >12 hours in past 4 weeks - PPO Visit: Rarely | 7 | 42
  Ring out for >12 hours in past 4 weeks - PPO Visit: Often | 0 | 2
  Ring out for >12 hours in past 4 weeks - PPO Visit: Missing | 6 | 13
  Ring out, even briefly, in past 4 weeks - Week 4 Visit: Never | 101 | 184
  Ring out, even briefly, in past 4 weeks - Week 4 Visit: Rarely | 1 | 11
  Ring out, even briefly, in past 4 weeks - Week 4 Visit: Often | 0 | 1
  Ring out, even briefly, in past 4 weeks - Week 4 Visit: Missing | 4 | 6
  Ring out, even briefly, in past 4 weeks - PPO Visit: Never | 91 | 121
  Ring out, even briefly, in past 4 weeks - PPO Visit: Rarely | 9 | 66
  Ring out, even briefly, in past 4 weeks - PPO Visit: Often | 0 | 2
  Ring out, even briefly, in past 4 weeks - PPO Visit: Missing | 6 | 13

15. Secondary Outcome: Acceptability: Participants Who Are Satisfied With the Study Products for Preventing HIV
Description: Based on participant report of how satisfied they have been with the the study product they were randomized to receive for HIV prevention. Only asked of participants in Cohorts 2 and 3.
Time Frame: Measured at Week 4 visits.
Population: Participants enrolled and randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Mothers: Truvada Tablet | Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Mothers: Truvada Tablet
Number analyzed (Participants) | 104 | 48 | 199 | 49
Participants
  Very satisfied | 68 | 27 | 125 | 25
  Satisfied | 34 | 17 | 73 | 22
  Neutral | 1 | 1 | 0 | 1
  Dissatisfied | 0 | 0 | 0 | 1
  Very dissatisfied | 0 | 0 | 0 | 0
  Missing | 1 | 3 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the duration of participants' time on study. For mothers, this ranged up to 36 weeks, depending on the participants' gestational age at enrollment and when their pregnancy outcome occurred. Adverse event data for mothers was collected up to 8 weeks after pregnancy outcome. For infants, their duration of time on study was 1 year.
Description: The "Any Event in SOC" rows summarize the total number of adverse events within an SOC. These events are also summarized using the specific Adverse Event Term for the event.
Groups:
- Cohort 1 Mothers: Dapivirine (DPV) Vaginal Ring (VR): Participants in Cohort 1 (36 0/7 weeks - 37 6/7 weeks) will use one DPV VR continuously for approximately one month, replacing the DPV VR each month. Participants will use the DPV VR until their pregnancy outcome but no later than 41 6/7 weeks of gestation.Dapivirine (DPV) Vaginal Ring (VR): Vaginal ring containing 25 mg of DPV
- Cohort 1 Mothers: Truvada Tablet: Participants in Cohort 1 (36 0/7 weeks - 37 6/7 weeks) will take one Truvada oral tablet daily. Participants will take Truvada until their pregnancy outcome but no later than 41 6/7 weeks of gestation.Truvada Tablet: Tablet taken orally
- Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR): Participants in Cohort 2 (30 0/7 weeks - 35 6/7 weeks) will use one DPV VR continuously for approximately one month, replacing the DPV VR each month. Participants will use the DPV VR until their pregnancy outcome but no later than 41 6/7 weeks of gestation.Dapivirine (DPV) Vaginal Ring (VR): Vaginal ring containing 25 mg of DPV
- Cohort 2 Mothers: Truvada Tablet; Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR): Participants in Cohort 2 (30 0/7 weeks - 35 6/7 weeks) will take one Truvada oral tablet daily. Participants will take Truvada until their pregnancy outcome but no later than 41 6/7 weeks of gestation.Truvada Tablet: Tablet taken orally
- Cohort 3 Mothers: Truvada Tablet: Participants in Cohort 3 (12 0/7 weeks - 29 6/7 weeks) will take one Truvada oral tablet daily. Participants will take Truvada until their pregnancy outcome but no later than 41 6/7 weeks of gestation.Truvada Tablet: Tablet taken orally
- Cohort 1 Infants: Dapivirine (DPV) Vaginal Ring (VR): Infants born to maternal participants in the Cohort 1 (36 0/7 weeks - 37 6/7 weeks) DPV VR arm.Dapivirine (DPV) Vaginal Ring (VR): Vaginal ring containing 25 mg of DPV
- Cohort 1 Infants: Truvada Tablet: Infants born to maternal participants in the Cohort 1 (36 0/7 weeks - 37 6/7 weeks) Truvada oral tablet daily arm.Truvada Tablet: Tablet taken orally
- Cohort 2 Infants: Dapivirine (DPV) Vaginal Ring (VR): Infants born to maternal participants in the Cohort 2 (30 0/7 weeks - 35 6/7 weeks) DPV VR arm.Dapivirine (DPV) Vaginal Ring (VR): Vaginal ring containing 25 mg of DPV
- Cohort 2 Infants: Truvada Tablet: Infants born to maternal participants in the Cohort 2 (30 0/7 weeks - 35 6/7 weeks) Truvada oral tablet daily arm.Truvada Tablet: Tablet taken orally
- Cohort 3 Infants: Dapivirine (DPV) Vaginal Ring (VR): Infants born to maternal participants in the Cohort 3 (12 0/7 weeks - 29 6/7 weeks) DPV VR arm.Dapivirine (DPV) Vaginal Ring (VR): Vaginal ring containing 25 mg of DPV
- Cohort 3 Infants: Truvada Tablet: Infants born to maternal participants in the Cohort 3 (12 0/7 weeks - 29 6/7 weeks) Truvada oral tablet daily arm.Truvada Tablet: Tablet taken orally
Arm/Group | Cohort 1 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 1 Mothers: Truvada Tablet | Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Mothers: Truvada Tablet | Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Mothers: Truvada Tablet | Cohort 1 Infants: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 1 Infants: Truvada Tablet | Cohort 2 Infants: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 2 Infants: Truvada Tablet | Cohort 3 Infants: Dapivirine (DPV) Vaginal Ring (VR) | Cohort 3 Infants: Truvada Tablet
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/49 | 0/106 | 0/51 | 0/202 | 0/49 | 0/99 | 1/48 | 4/103 | 0/51 | 4/197 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/101 | 3/49 | 8/106 | 2/51 | 11/202 | 2/49 | 14/99 | 7/48 | 22/103 | 5/51 | 30/197 | 3/48
Other Adverse Events (participants affected / at risk) | 43/101 | 29/49 | 73/106 | 39/51 | 169/202 | 37/49 | 91/99 | 39/48 | 92/103 | 44/51 | 176/197 | 43/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Mothers: Dapivirine (DPV) Vaginal Ring (VR) (N=101) | Cohort 1 Mothers: Truvada Tablet (N=49) | Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) (N=106) | Cohort 2 Mothers: Truvada Tablet (N=51) | Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR) (N=202) | Cohort 3 Mothers: Truvada Tablet (N=49) | Cohort 1 Infants: Dapivirine (DPV) Vaginal Ring (VR) (N=99) | Cohort 1 Infants: Truvada Tablet (N=48) | Cohort 2 Infants: Dapivirine (DPV) Vaginal Ring (VR) (N=103) | Cohort 2 Infants: Truvada Tablet (N=51) | Cohort 3 Infants: Dapivirine (DPV) Vaginal Ring (VR) (N=197) | Cohort 3 Infants: Truvada Tablet (N=48)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital absence of bile ducts (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmorphism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pectus excavatum (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trisomy 21 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden infant death syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amniotic cavity infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 4 (4) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Neonatal pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 4 (5) | 1 (1) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Neonatal hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Placenta praevia haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary haemosiderosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Mothers: Dapivirine (DPV) Vaginal Ring (VR) (N=101) | Cohort 1 Mothers: Truvada Tablet (N=49) | Cohort 2 Mothers: Dapivirine (DPV) Vaginal Ring (VR) (N=106) | Cohort 2 Mothers: Truvada Tablet (N=51) | Cohort 3 Mothers: Dapivirine (DPV) Vaginal Ring (VR) (N=202) | Cohort 3 Mothers: Truvada Tablet (N=49) | Cohort 1 Infants: Dapivirine (DPV) Vaginal Ring (VR) (N=99) | Cohort 1 Infants: Truvada Tablet (N=48) | Cohort 2 Infants: Dapivirine (DPV) Vaginal Ring (VR) (N=103) | Cohort 2 Infants: Truvada Tablet (N=51) | Cohort 3 Infants: Dapivirine (DPV) Vaginal Ring (VR) (N=197) | Cohort 3 Infants: Truvada Tablet (N=48)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 12 (12) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Birth mark (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Congenital absence of bile ducts (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital inguinal hernia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 7 (7) | 1 (1)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macrocephaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail aplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polydactyly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tethered oral tissue (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinopathy of prematurity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal skin tags (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 6 (6) | 7 (7) | 9 (9) | 2 (2) | 15 (15) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 14 (14) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infantile colic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 8 (8) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 9 (9) | 0 (0) | 6 (6) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Developmental delay (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 4 (4) | 1 (1) | 5 (5) | 2 (2)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess of eyelid (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amoebiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amoebic dysentery (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bullous impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 4 (4) | 2 (2) | 12 (12) | 4 (4)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 8 (8) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatophytosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 11 (11) | 1 (1) | 15 (15) | 7 (7) | 26 (26) | 13 (13) | 52 (52) | 14 (14)
Genitourinary chlamydia infection (Infections and infestations) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 8 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genitourinary tract gonococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Giardiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hookworm infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 5 (5) | 1 (1)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 8 (8) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 4 (4) | 1 (1) | 5 (5) | 0 (0)
Malaria (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 3 (3) | 3 (3) | 3 (3)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 7 (7) | 1 (1)
Ophthalmia neonatorum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 15 (15) | 4 (4)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 4 (4)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 4 (4) | 1 (1) | 21 (21) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postpartum sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Schistosomiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea capitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2) | 12 (12) | 7 (7) | 36 (36) | 7 (7) | 54 (54) | 23 (23) | 62 (62) | 33 (33) | 127 (127) | 24 (24)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 9 (9) | 5 (5) | 12 (12) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0) | 8 (8) | 0 (0) | 13 (13) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginitis trichomonal (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foreign body in ear (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyphaema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site discharge (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Uterine cervical laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 5 (5) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 2 (2) | 1 (1) | 6 (6) | 3 (3) | 20 (20) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 7 (7) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 6 (6) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Feeding disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 34 (34) | 16 (16) | 45 (45) | 14 (14) | 48 (48) | 11 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 8 (8) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 2 (2) | 6 (6) | 4 (4) | 12 (12) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 10 (10) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Caput succedaneum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 2 (2) | 4 (4) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
False labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 11 (11) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2) | 5 (5) | 6 (6) | 16 (16) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intrapartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 10 (10) | 5 (5) | 8 (8) | 4 (4)
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructed labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post abortion haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 5 (5) | 4 (4) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 15 (15) | 9 (9) | 29 (29) | 13 (13) | 51 (51) | 10 (10)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perinatal depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ketonuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 12 (12) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral perforation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lactation insufficiency (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nipple disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic organ prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 10 (10) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 8 (8) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 3 (3) | 6 (6) | 2 (2) | 7 (7) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 2 (2) | 3 (3) | 6 (6) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 6 (6) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 5 (5) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pityriasis alba (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient neonatal pustular melanosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical discharge (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT03965923/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT03965923/SAP_002.pdf